CLINICAL TRIAL: NCT03676127
Title: Diagnostic Accuracy of Between Side Differences of Ultrasonographic Dermal Thickness Measurements in Breast Cancer Related Arm Lymphedema
Brief Title: Diagnostic Accuracy of Dermal Thickness in Lymphedema
Status: Completed | Type: Observational
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Other Study IDs: 09.2018.
Record Dates: First submitted 2018-09-16; First posted 2018-09-18 (Actual); Last update posted 2018-12-20 (Actual); Status verified 2018-12

CONDITIONS: Lymphedema of Upper Arm; Breast Cancer
Keywords: assessment; breast cancer; diagnosis; lymphedema; measurement; ultrasound
MeSH Terms: conditions — Breast Neoplasms; Disease; Lymphedema

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study Group: ultrasonographic dermal thickness measurements in patients with unilateral breast cancer related lymphedema
  Interventions: Other: ultrasonographic dermal thickness measurements

INTERVENTIONS:
Other: ultrasonographic dermal thickness measurements — ultrasonographic dermal thickness measurements

SUMMARY:
Ultrasound is an easily feasible noninvasive technique which is widely used in rehabilitation settings. Measurement of dermal thickness via ultrasound can be less time consuming than volume measurements with water displacement and circumference measurements. Measurement of subcutaneous tissue thickness were used for both assessment and treatment outcome. Recently reliability of ultrasound examination of thickness of the skin and subcutaneous tissue were studied by Han et al. However, diagnostic accuracy of this method has not been studied before. Early identification of breast cancer related lymphedema to start treatment earlier is critical. Consequently, reliability and diagnostic accuracy of the assessment techniques of lymphedema is crucial to evaluate both severity at the time of diagnosis, and later effectiveness of treatment. The aim of this study was to establish diagnostic accuracy of between side differences of ultrasonographic dermal thickness measurements in breast cancer related arm lymphedema.

DETAILED DESCRIPTION:
Breast cancer related arm lymphedema is a potential sequalae from the treatment of breast cancer which is characterized by the accumulation of protein-rich lymphatic fluid in the extracellular spaces. It may occur in almost 40% of the patients who have undergone breast cancer surgery or radiation therapy. Breast cancer related lymphedema may appear in the upper extremity, as well as in the ipsilateral upper quadrant and remaining breast tissue. Clinically, the diagnosis of lymphedema is based mainly on patient history and self-report of symptoms, visual inspection and skin palpation, and the determination of volume differences between both limbs. The most widely accepted measure of lymphedema is limb volume compared with that of the unaffected limb or compared with that of the same limb. Sequential circumference measurements along designated measure points are widely used in clinical practice. Limb volumes can be calculated or estimated based on a truncated cone formula. Volumetry by means of water displacement is considered the golden standard. The most common criterion for lymphedema diagnosis is a volume difference of 200 mL. Circumference measurements and the estimated volume were found to be reliable and highly correlated with each other. However, these volume measurements are not only influenced by fluid changes but also by compositional changes of muscle mass, bone, or fat. Also, water displacement is too cumbersome and messy to be used in routine clinical practice.

Ultrasound is an easily feasible noninvasive technique which is widely used in rehabilitation settings. Measurement of dermal thickness via ultrasound can be less time consuming than volume measurements with water displacement and circumference measurements. Measurement of subcutaneous tissue thickness were used for both assessment and treatment outcome. Recently reliability of ultrasound examination of thickness of the skin and subcutaneous tissue were studied by Han et al. However, diagnostic accuracy of this method has not been studied before. Early identification of breast cancer related lymphedema to start treatment earlier is critical. Consequently, reliability and diagnostic accuracy of the assessment techniques of lymphedema is crucial to evaluate both severity at the time of diagnosis, and later effectiveness of treatment. The aim of this study was to establish diagnostic accuracy of between side differences of ultrasonographic dermal thickness measurements in breast cancer related arm lymphedema. Patients with breast cancer related lymphedema will be included. Lymphedema of the limbs will be assessed using the circumferential method. The circumferential upper limb measurementswill be carried out with the arm abducted at 30°, starting at the level of the carpometacarpal joint, every 5 cm proximal to this point along both limbs. Then, a computer program (limb volumes professional version 5.0) will be used to convert these values into limb volumes in milliliters. Differences in volume of affected and unaffected sides was defined as edema (volume difference). The criterion for lymphedema diagnosis is volume difference of 200 mL. Ultrasonographic dermal thickness measurements will be performed from medial forearm. Differences of the affected and unaffected sides will be calculated. The circumference measurement method and the thickness of the skin of the edematous limb by using the ultrasound and the truncated cone method by using circumference measurements will be compared to evaluate the diagnostic accuracy of between side differences of ultrasonographic dermal thickness measurements in breast cancer related arm lymphedema.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with unilateral postmastectomy lymphedema

Exclusion Criteria:

1. Bilateral lymphedema
2. The patients who had known systemic edemagenic conditions (e.g., cardiac/hepatic/renal failure, terminal cancer, on chemotherapy), and/or with cancer recurrence

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with breast cancer related lymphedema
Sampling Method: Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2018-09-28 (Actual); Primary Completion 2018-12-19 (Actual); Study Completion 2018-12-19 (Actual)

PRIMARY OUTCOMES:
Area under curve | Day 0
  Area under curve

SECONDARY OUTCOMES:
Sensivity of between side differences of ultrasonographic dermal thickness measurements | Day 0
  Sensivity of between side differences of ultrasonographic dermal thickness measurements
Specificity of between side differences of ultrasonographic dermal thickness measurements | Day 0
  Specificity of between side differences of ultrasonographic dermal thickness measurements
Interlimb volume difference | Day 0
  Interlimb volume differencedetected via truncated cone method from circumference measurements
between side differences of ultrasonographic dermal thickness measurements | Day 0
  between side differences of ultrasonographic dermal thickness measurements

CONTACTS AND LOCATIONS:
Overall Officials: Esra Giray, MD, Principal Investigator — Marmara University
Locations (1):
- Esra Giray, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The investigators don't plan to share IPD.

REFERENCES:
- [Background] Yang EJ, Kim SY, Lee WH, Lim JY, Lee J. Diagnostic Accuracy of Clinical Measures Considering Segmental Tissue Composition and Volume Changes of Breast Cancer-Related Lymphedema. Lymphat Res Biol. 2018 Aug;16(4):368-376. doi: 10.1089/lrb.2017.0047. Epub 2018 Jan 17. PMID 29338541
- [Background] Tassenoy A, De Strijcker D, Adriaenssens N, Lievens P. The Use of Noninvasive Imaging Techniques in the Assessment of Secondary Lymphedema Tissue Changes as Part of Staging Lymphedema. Lymphat Res Biol. 2016 Sep;14(3):127-33. doi: 10.1089/lrb.2016.0011. PMID 27631582
- [Background] Suehiro K, Morikage N, Yamashita O, Harada T, Samura M, Takeuchi Y, Mizoguchi T, Nakamura K, Hamano K. Skin and Subcutaneous Tissue Ultrasonography Features in Breast Cancer-Related Lymphedema. Ann Vasc Dis. 2016;9(4):312-316. doi: 10.3400/avd.oa.16-00086. Epub 2016 Nov 25. PMID 28018504
- [Background] Bok SK, Jeon Y, Hwang PS. Ultrasonographic Evaluation of the Effects of Progressive Resistive Exercise in Breast Cancer-Related Lymphedema. Lymphat Res Biol. 2016 Mar;14(1):18-24. doi: 10.1089/lrb.2015.0021. Epub 2016 Jan 29. PMID 26824517
- [Background] Han N, Cho Y, Hwang J, Kim H, Cho G. Usefulness of ultrasound examination in evaluation of breast cancer-related lymphedema. J Korean Acad Rehabil Med. 2011;35:101-9.